CLINICAL TRIAL: NCT01313806
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study to Evaluate the Efficacy of the Application of Magnetic Fields Using the Resonator for the Treatment of Alzheimer"s Disease in Addition to Standard of Care
Brief Title: Study of Magnetic Fields to Treat Alzheimer's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: pico-tesla Magnetic Therapies, LLC (Industry)
Responsible Party: Allen S. Braswell CEO, pico-tesla Magnetic Therapies, LLC, Pico-Tesla Magnetic Therapies, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WIRB 1123661
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Alzheimer's Disease
Keywords: dementia; memory loss; cognitive decline
MeSH Terms: conditions — Alzheimer Disease; Dementia; Memory Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resonator (Active Comparator): Treatment with active Resonator device using low level magnetic fields
  Interventions: Device: Resonator
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Resonator — Treatment group vs. Placebo group
  Arms: Resonator
Device: Placebo — Inactive Resonator Device
  Arms: Placebo

SUMMARY:
To determine if low level magnetic fields can help to improve memory in patients diagnosed with Alzheimer's disease.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine whether application of magnetic fields generated by the Resonator may improve cognitive functioning and memory in individuals with a diagnosis of Alzheimer"s dementia, as an adjunctive therapy to standard of care.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for participation in this clinical study, a subject must satisfy each of the following "Inclusive Conditions" criteria.

* Current diagnosis of Alzheimer's Disease appropriately documented by the patients physician and/or neurologist
* Documentation verifying that other generally recognized causes of dementia have been ruled out by prior physician evaluations
* Mild to Moderate Dementia, as evidenced by a score of not less than 12 nor greater than 26 on the Mini Mental Status Exam (MMSE).
* Subject is ambulatory
* A Study Partner who can attend all study visits with the subject. Study Partner being defined as an adult who has at least 10 hours/week of contact with the subject, and can accompany the subject to all testing and treatment study visits.
* Stable "anti-dementia" medication regimen without significant side effects for at least 3 months, and on stable medication (unrelated to anti-dementia) without significant side effects for at least 1 month; willingness and ability to maintain the stable medication regimen throughout the course of the study.
* Willingness and ability to present to the testing center for all study evaluations
* Willingness and ability to present to the treatment center for all study treatments (exposure to the Resonator™)
* Willingness to maintain stable diet and activity regimen for the duration of the study.
* Willing and able to abstain from partaking in any non-essential (not physician ordered) existing or new treatments to improve cognition and mental functioning
* Willing and able to abstain from any medications that could affect cognition and mental functioning during the course of the study
* Male or female.
* Any ethnic background.
* Age 55 and older.

Exclusion Criteria A subject will be considered ineligible for participation in this clinical study if he or she satisfies any one or more of the following exclusive conditions criteria.

* Change in anti-dementia medical regimen within 3 months prior to initiation of study.
* Confirmed diagnosis other non-Alzheimer's type of dementia
* Significant neurologic or psychiatric illness other than Alzheimer's disease
* Unstable cardiac disease, such as any history of cardiac arrhythmias (including atrial fibrillation, ventricular fibrillation, or irregular atrial-ventricular conduction time), or any incidences of congestive heart failure, or myocardial infarction, within the last six months.
* Previous surgical interventions involving prosthetics or implants comprised of ferrous metals, or pacemakers, vagus nerve stimulators, or other functional electrical stimulators such as those commonly used for pain.
* Reported consumption of more than 14 alcoholic drinks per week.
* Uncontrolled hypertension.
* Uncontrolled atrial fibrillation or other uncontrolled arrhythmias, e.g. tachycardia, bradycardia.
* Uncontrolled seizure disorder.
* History of seizures or usage of anti-seizure medications that, in the opinion of the investigator, participation in this trial would represent a risk to the subject.
* Uncontrolled, unstable, or untreated medical conditions which may significantly impact the subject's health or ability to complete the entire study, in the opinion of the investigator.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cog (ADAS-cog) | end of treatment at 12 weeks

SECONDARY OUTCOMES:
Mini-Mental Status Exam (MMSE), Neuropsychiatric Inventory Questionnaire (NPI-Q), Clinical Dementia Scale | end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Klapper, MD, Principal Investigator — Mile High Research Center; Miguel Trevino, MD, Principal Investigator — Innovative Research of West Florida
Locations (2):
- United States (2):
  - Mile High Research Center, Denver, Colorado
  - Innovative Research of West Florida, Clearwater, Florida